CLINICAL TRIAL: NCT06495957
Title: Evaluation of Therapeutic Effect and Brain Mechanism of Electroacupuncture in Treating Agitation Symptoms of Alzheimer's Disease
Brief Title: Electroacupuncture for the Treatment of Agitated Symptoms of Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Bao-Hui Jia, Director of rehabilitation Medicine, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-075-KY-01
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Agitation Associated With Alzheimer's Dementia; Alzheimer's Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Needles will be inserted at 11 acupoints. Acupoints will be added electrical stimulation via a low-frequency neural regulator (electrical stimulator) respectively with a disperse-dense wave after insertion of all needles. Twenty-minute treatments will be delivered three times weekly for 8 weeks.
  Interventions: Other: Electroacupuncture group
- Micro-acupuncture group (Other): 11 needles will be inserted at acupoints with 1-3 mm in depth. The acupoints will then be connected to the electrical stimulator in accordance with the electroacupuncture group. The frequency of the electroacupuncture is the same as that of the electroacupuncture group, which is briefly energized at the beginning for 30s.Twenty-minute treatments will be delivered three times weekly for 8 weeks.
  Interventions: Other: Micro-acupuncture group

INTERVENTIONS:
Other: Electroacupuncture group — Electroacupuncture treatment consists of conventional acupuncture and electrical stimulation. After acupuncture, the electrical stimulation is continuously stimulated for 20 minutes.
  Arms: Electroacupuncture group
Other: Micro-acupuncture group — After acupuncture, the electrical stimulation is continuously stimulated for 20 minutes. Electrical stimulation is applied briefly for the first 30 seconds.
  Arms: Micro-acupuncture group

SUMMARY:
The purpose of this study is to evaluate the efficacy of electroacupuncture in the treatment of agitation symptoms in patients with Alzheimer's disease (AD). Meanwhile the study aims to explore the brain central mechanism of electroacupuncture in the treatment of agitation symptoms in patients with AD by using resting state functional magnetic resonance technology.

DETAILED DESCRIPTION:
This is a multicenter, parallel-group, patient-blinded and outcome-assessor-blinded randomized controlled trial consisting of two stages: a 8-week treatment period followed by a 8-week follow-up period. The study aims to assess therapeutic efficacy and safety of electroacupuncture for agitated symptoms of AD. Approximately 224 AD patients with symptoms of agitation will be randomly assigned to the electroacupuncture group or micro-electroacupuncture group. 50 patients in each of the two groups will be selected to complete rs-fMRI scans before the initial treatment and after the last treatment in order to investigate the central mechanism underlying the effects of electroacupuncture treatment on functional activity in patients with AD patients with symptoms of agitation.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the revised draft diagnostic criteria for Alzheimer's disease published by the Alzheimer's Association in 2023
2. Meet the 2023 IPA definition of agitated symptoms of cognitive impairment
3. Cohen Mansfield Agitation Inventory (CMAI)≥45 points
4. Have been on stable anti-AD medication (cholinesterase inhibitors, etc.) for more than 1 month
5. If taking antipsychotics, the medication regimen for agitation (antipsychotics) is stable for 1 month prior to randomization
6. Subject and legal guardian and caregiver sign informed consent.

Exclusion Criteria:

1. There are contraindications for acupuncture treatment, such as the tendency of acupoint bleeding or allergy to metal
2. Received electroacupuncture treatment in the past 2 weeks
3. At the time of the screening, participants are participating in other clinical trials or planned to participate in other clinical trials in the next 17 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Cohen Mansfield Agitation Inventory (CMAI) | CMAI will be evaluated after the final treatment at week 8
  CMAI is one of the most widely used tools for assessing agitated behaviors that affect patients' quality of life and burden caregivers. The scale contains 29 items, including different agitated behaviors and emotional states, to which the assessed responds based on their own observations and experiences. The scores for all items are added together to give a total score. The higher the score, the more severe the agitated behavior.

SECONDARY OUTCOMES:
Cohen Mansfield Agitation Inventory (CMAI) | The CMAI will be evaluated at week 4 of treatment and at week 4 and week 8 of follow-up
  CMAI is one of the most widely used tools for assessing agitated behaviors that affect patients' quality of life and burden caregivers. The scale contains 29 items, including different agitated behaviors and emotional states, to which the assessed responds based on their own observations and experiences. The scores for all items are added together to give a total score. The higher the score, the more severe the agitated behavior.
Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change(mADCS-CGIC) | The mADCS-CGIC assessment will be completed before treatment and at week 8 of treatment.
  mADCS-CGIC is a global rating of change developed to assess clinically significant change in symptoms over time in AD clinical trials. Clinicians rate patient agitation on the mADCS-CGIC as: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), and very much worse (7) compared to baseline symptoms.
the Behavioral Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) | The BEHAVE-AD assessment will be completed before treatment and at week 8 of treatment.
  The BEHAVE-AD scale is used to assess the behavioral pathology of patients with Alzheimer's disease. It contains 25 items to assess patients' symptoms and severity across multiple behavioral areas. The higher the total score of BEHAVE-AD, the more serious the behavioral pathology of the patient.
Neuropsychiatric Inventory (NPI) | NPI will be completed before treatment and at week 8 of treatment.
  NPI is used to evaluate neuropsychiatric behavioral symptoms of dementia patients. The scale assesses the neuropsychiatric disorders of patients according to the caregiver's view of the patient's behavior and the corresponding distress felt by the patient. The scoring range of the patient evaluation scale is 0-144 points, and the scoring of the caregiver distress scale is 0-60 points, the lower the score is, the better the patient's condition is.
Mini-mental State Examination (MMSE) | MMSE will be completed before treatment and at week 8 of treatment.
  The MMSE scale can comprehensively, accurately and quickly reflect the intellectual state and cognitive function defect of the subjects. The total score ranges from 0 to 30 points, and the higher the score is, the better the cognitive function is
Alzheimer disease assessment scale cognition (ADAS-Cog) | ADAS-Cog scale will be completed before treatment and at week 8 of treatment.
  The ADAS-Cog scale is a scale commonly used to assess cognitive impairment in Alzheimer's patients on a scale ranging from 0 to 70 points, with higher scores indicating more severe cognitive impairment.
Activities of daily living (ADL) | ADL scale will be completed before treatment and at week 8 of treatment.
  The ADL consists of the Physical self-maintenance scale (PSMS) and the Instrumental Activities of daily living Scale (IADL). Higher scores indicating lower ability.
Pittsburgh Sleep Quality Index (PSQI) | PSQI will be completed before treatment and at week 8 of treatment.
  The PSQI Scale is a standardized tool used to assess sleep quality and contains 7 sections covering the main aspects of sleep quality. Each section was scored on a scale of 0-3, and the overall score was 0-21, with higher scores indicating poorer sleep quality.
Zarit Burden Interview(ZBI) | ZBI will be completed before treatment and at week 8 of treatment.
  The ZBI scale is a tool used to assess the degree of psychological and physical burden on caregivers caring for family members with cognitive impairment or chronic illness. The total score ranges from 0 to 88, with higher scores indicating higher caregiving burden.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Jia, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (7):
- China (7):
  - Beijing United Family Rehabilitation Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Geriatric Hospital, Beijing, Beijing Municipality
  - Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No